CLINICAL TRIAL: NCT00001651
Title: Studies of Lymphocyte Kinetics Using Stable Isotopes
Brief Title: Use of Labeled Glucose to Study Lymphocyte Replication and Survival in HIV-Infected Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow/Insufficient accrual
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 970191; 97-I-0191
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: HIV; Healthy Volunteers
Keywords: HIV Infection; Lymphocyte Turnover
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: [6,6-2H2]-glucose will be administered as a continuous IV infusion for one to five days. Blood (approximately 30-50 ml) will be drawn every one to three days during the infusion to obtain cells for analysis. In addition, serum glucose will be checked every two to three days. Following completion of the infusion, blood may be drawn daily for the first week, and then twice weekly for an additional 3 weeks, and then weekly to monthly.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIV-infected subjects (Experimental): HIV-infected adults
  Interventions: Other: [6,6-2H2]-glucose
- HIV-negative subjects (Experimental): HIV-negative adults
  Interventions: Other: [6,6-2H2]-glucose

INTERVENTIONS:
Other: [6,6-2H2]-glucose — [6,6-2H2]-glucose will be administered as a continuous IV infusion for one to five days.

SUMMARY:
This study will examine how quickly white blood cells called CD4 lymphocytes replicate (divide) and how long they live in both HIV-infected and non-infected people by measuring how quickly the genetic material (DNA) of cells is replicated. To do this, participants will receive infusions of glucose, a non-radioactive form of a type of sugar. Cells normally use glucose to make various products needed for cell growth and replication, including cell DNA. Measuring how much glucose cells incorporate into their DNA can provide important information about cell replication. This rate of incorporation will be examined and compared in HIV-infected people and in healthy, normal volunteers.

HIV-infected patients and non-infected healthy volunteers 18 years of age and older may be eligible for this study. Candidates will be screened with a medical history, physical examination, chest X-ray, electrocardiogram (EKG) and blood tests.

Participants will be given a continuous infusion of glucose at a dose of up to 60 grams (about 2 ounces) per day for up to 5 days. The glucose will be delivered through a catheter (thin plastic tube) placed in an arm vein. Blood samples will be collected as often as daily in the first week following the infusion and then from twice a week to once a month for up to 4 years. Alternatively, patients may undergo leukapheresis a procedure for collecting quantities of lymphocytes up to 10 times during the first month after the infusion, and possibly later as well, but no more often than once every 2 weeks. For this procedure, whole blood is collected through a needle in an arm vein. The blood circulates through a machine that separates it into its components. The white cells are removed and the rest of the blood is returned to the body either through the same needle or through a second needle in the other arm. Participants may be asked to receive up to four glucose infusions. There will be at least a 2-week interval between infusions. Participants who have more than three leukapheresis procedures within 3 weeks will have at least 6 weeks between infusions.

Participants will be followed periodically in the outpatient clinic for evaluation and tests.

This study may provide a better understanding of how HIV causes disease and progressive weakening of the immune system and how therapies affect immunity.

DETAILED DESCRIPTION:
Understanding the rate of lymphocyte replication and destruction in HIV-infected patients, as well as the effects of therapy on lymphocyte replication should lead to a better understanding of the mechanisms behind the immunodeficiency induced by HIV. To examine this directly, up to 100 HIV-infected patients will receive up to 5 days of continuous infusions with [6,6-(2)H(2)]-glucose, a nonradioactive, stable isotope of glucose that is safe to administer. The deuterium is incorporated into DNA via metabolism of glucose to ribose and incorporation into nucleotides. The rate of incorporation can be measured in subpopulations of cells to determine the rate of replication of those cells. Fifty HIV-uninfected persons will also be enrolled in the protocol to allow a determination of lymphocyte kinetics in individuals with normally functioning immune systems or immune systems that may have been affected by other diseases. All participants in this study will be reimbursed for the inconvenience and discomfort associated with study participation.

ELIGIBILITY:
* INCLUSION CRITERIA:

FOR PATIENTS:

18 years or older.

Able to provide informed consent and willing to comply with study requirements and clinic policies.

Negative urine pregnancy test (for women of childbearing potential).

Hemoglobin greater than 10 mg/dl.

Adequate venous access in the arms for blood drawing and 5 day infusions, and lymphapheresis

Willingness to allow stored samples to be used for future studies of HIV infection and/or immunological function, and willingness to have HLA typing performed. (For previously enrolled patients, patients would be requested, but not required, to provide permission to use stored samples in the future, and to permit HLA testing

FOR HIV POSITIVE PATIENTS:

Documented HIV infection (ELISA/Western blot positive or, for acute seroconverters, PCR positive).

FOR HIV NEGATIVE PATIENTS:

Negative ELISA/Western blot.

EXCLUSION CRITERIA:

Diabetes mellitus requiring drug therapy.

Active substance abuse or prior history of substance abuse which may interfere with protocol compliance.

Psychiatric illness or disturbance which, in the assessment of the protocol team, may affect patient safety or compliance.

Significant underlying cardiac, pulmonary, renal, gastrointestinal, rheumatologic or CNS disease as detectable on routine history, physical exam, or screening laboratory studies. Patients would be excluded if they had an acute or chronic underlying medical problem that in the judgment of the principal investigator could be exacerbated by participating in the protocol or that would make it difficult for them to comply with the protocol requirements.

Pregnancy or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 1998-02-25 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-05-29 (Actual)

PRIMARY OUTCOMES:
Kinetics of lymphocyte turnover | Day 2, 5 (end of [6,6-2H2]-glucose infusion), 6, 8, 12, 16, 20, and 28. After day 28, visits will occur monthly through 6 months, then no more often than every 3 months through 2 years.
  Cell turnover markers

CONTACTS AND LOCATIONS:
Overall Officials: Joseph A Kovacs, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Wolthers KC, Bea G, Wisman A, Otto SA, de Roda Husman AM, Schaft N, de Wolf F, Goudsmit J, Coutinho RA, van der Zee AG, Meyaard L, Miedema F. T cell telomere length in HIV-1 infection: no evidence for increased CD4+ T cell turnover. Science. 1996 Nov 29;274(5292):1543-7. doi: 10.1126/science.274.5292.1543. PMID 8929418
- [Background] Ho DD, Neumann AU, Perelson AS, Chen W, Leonard JM, Markowitz M. Rapid turnover of plasma virions and CD4 lymphocytes in HIV-1 infection. Nature. 1995 Jan 12;373(6510):123-6. doi: 10.1038/373123a0. PMID 7816094
- [Background] Hellerstein MK. Methods for measurement of fatty acid and cholesterol metabolism. Curr Opin Lipidol. 1995 Jun;6(3):172-81. doi: 10.1097/00041433-199506000-00010. PMID 7648007
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1997-I-0191.html